CLINICAL TRIAL: NCT04262063
Title: Effectiveness of Tell Play do Technique in Comparison to Tell Show do Technique for the Management of Anxious Children: A Randomized Controlled Trial
Brief Title: Effectiveness of TPD Tech VS TSD Tech
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: rehab abdulhameed ebrahim mohammed (Other)
Responsible Party: Sponsor-Investigator, rehab abdulhameed ebrahim mohammed, principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eff of TPD vsTSD
Record Dates: First submitted 2020-02-02; First posted 2020-02-10 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Dental Anxiety
Keywords: tell show do; tell play do; dental anxiety; child behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: parallel group two arms superiority trial with 1:1 allocation ratio
Who Masked: Participant
Masking Description: The patients, their parents and the statistician will be blinded ,
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tell play do technique (Experimental): Tell play do technique with a dental imitation toy and using euphemisms instead of demonstrating on a model or observing one. Tell play do technique provides a better explanatory concept of the dental procedure and can lead to more cooperation of the children patients which can influence the dental treatment in a good and positive way.
  Interventions: Behavioral: Tell play do technique
- tell show do technique (Active Comparator): Tell show do is the gold standard of the non-pharmacological behavior management techniques. It is based on the principle of learning theory and it is performed by the dentists themselves . It is the most important behavior modification technique practiced by dentists and it is commonly used for management of children anxiety in the first dental visit .
  Interventions: Behavioral: tell show do

INTERVENTIONS:
Behavioral: Tell play do technique — it apply the concept of learning by doing .children will enjoy playing with customized dental models
  Arms: tell play do technique
Behavioral: tell show do — Tell: your dentist explaining to you what they'd like to do Show: showing you what is involved (e. g. showing the equipment and demonstrating it on a finger) Do: performing the procedure
  Arms: tell show do technique

SUMMARY:
Assessment of the effectiveness of tell play do technique and tell show do technique in management of anxious children .

DETAILED DESCRIPTION:
Child dental anxiety has been a matter of concern for many years. It is defined as a nonspecific feeling of apprehension, worry, uneasiness and the source may be not clear or unknown .

Dental anxiety is considered as a major obstacle for the dental treatment. The dental appointment is a stressful situation specially for children which raises their anxiety level. Different studies among 6-12 years old children showed that 20%- 43 % exhibited high dental fear and anxiety .

Dental fear and anxiety can have negative implications for children's oral health. There is certainty for the negative impact of dental anxiety on the oral health-related quality of life of children, and studies have shown that children with dental fear and anxiety have worse oral health status than their peers (more untreated carious lesions).

It is also children with dental fear and anxiety may present with behavioral management problems which can disrupt the provision of dental treatment and negatively impact on the dental treatment the child receives. The anxiety experienced by children is not only distressing for the child, but it can also be a potentially stressful and upsetting experience for their parents .

A good patient-dentist relationship is crucial for the management of anxiety. It is the responsibility of pedodontists to make dentistry as child-friendly and pain-free as possible to bring about positive changes in the behavior of children during dental treatment .

Tell-show-do technique is widely used for managing pediatric dental patients. It is useful for almost all patients who can communicate, especially those patients who are 'monitors. Although widely used, the ability of this technique to prepare, and reduce child anxiety remains an area for research, because it's not always appropriate for those patients who are 'blunters' where detailed information can result in increased levels of anxiety .

So different modifications of this technique were used one of them is tell play do technique with a dental imitation toy and using euphemisms instead of demonstrating on a model or observing one. Tell play do technique provides a better explanatory concept of the dental procedure and can lead to more cooperation of the children patients which can influence the dental treatment in a good and positive way.

ELIGIBILITY:
Inclusion Criteria:

1. Children with Frankl's behavior rating score of 1,2 .
2. Patients with no previous dental experience.
3. Patients not suffering from cognitive or mental problems.
4. Children with primary molars indicated for extraction .
5. Age 4- 6 years old .

Exclusion Criteria:

1. Medically compromised patients
2. Patients suffering from cognitive or mental problems
3. Patients with previous dental experience

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
level of anxiety | Immediate In the first visit
  The level of dental anxiety of each patient will be assessed using finger pulse oximeter.

SECONDARY OUTCOMES:
change in behavior | immediate after the behavior management
  the operator will grade the child's behavior during the procedure using the (Face, Leg, Activity, Cry, Consolability) behavioral pain assessment scale.(FLACC)
  each category scores from 0-2 scale which result in a total score of 0-10
  0 relaxed and comfortable 1-3 mild discomfort 4-6 moderate pain 7-10 severe discomfort of pain or both
Ease of handling patients | immediate the end of the treatment
  The ease of handling the patient will be assessed using a validated questionnaire by 5-point Likert scale (1- Strong positive , 2- Positive, 3- Neutral , 4- Negative,5- Strong negative)
Ease of doing the procedures | immediate at the end of the treatment
  the ease of doing the procedures will be assessed using a validated questionnaire by 5-point Likert scale (1- Strong positive , 2- Positive, 3- Neutral , 4- Negative, 5- Strong negative)

IPD SHARING:
Plan to Share IPD: No